CLINICAL TRIAL: NCT03394443
Title: Which Needs for Premature New-born Babies' Parents Facing Environmental and Social Difficulties ? A Qualitative Study in Besancon University Hospital.
Brief Title: Which Needs for Premature New-born Babies' Parents Facing Environmental and Social Difficulties ?
Acronym: PrémaSoin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/347
Record Dates: First submitted 2017-12-28; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Semi-structured interviews — Semi-structured interviews of the parents of preterm infants. 3 weeks after their child has left hospital. They will be made either at the University Hospital of Besançon. They will take place in a dedicated hospital ward to ensure the confidentiality of the statements made between the investigator and the parent.
  They will follow a predefined questionnaire. They will be fully recorded on a dictaphone with note taking during the interview by the investigator and will be transcribed in writing anonymously and confidentially on Word.
  The content of the interviews will be analyzed:
  * As a first step, it will be a vertical analysis of the thematization of each interview
  * Then, in a second step, a transversal analysis between the contents of the different interviews.

SUMMARY:
This study aims to understand parents' needs regarding social difficulties faced in a child's preterm birth context.

DETAILED DESCRIPTION:
* From parents collected during semi-structured interviews.
* To highlight the social, environmental and economic difficulties that parents have encountered in the context of the premature birth of their child (before birth, during hospitalization and return home).
* Determine the possible help they need in the psychosocial and environmental field.
* Difficulties of the parents we expected:

  * Pre-existing child birth: poor socio-economic environment, unstable social, family and / or occupational status, poorly followed pregnancy, etc.
  * After the birth: professional break-up, custody of other children of the siblings, balance of the couple, financial loss, isolation, transportation problems to get to the hospital, etc.
* Needs we expected :

  * Before birth: measures to prevent prematurity, social and/or psychological support, information, etc.
  * After the birth: support of the entourage, interview with a social worker, help to come in hospital, help to live near the hospital, parental leave, project and long-term support, doctor referred, relationship with professionals in ambulatory (psychologist, Infant and Maternal Protection ...), preparation of the arrival of the child at home +/- home improvement, etc.

ELIGIBILITY:
Inclusion Criteria:

* Parents (father or mother ) of a premature new-born baby (< 37 SA) hospitalised in Besancon University Hospital at birth.

Exclusion Criteria:

* Parents < 18 years old
* Refusing to participate

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of a premature new-born baby (< 37 SA)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Social, environmental and economic difficulties encountered by parents | Month 1
  Qualitative analysis of semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No